CLINICAL TRIAL: NCT03129815
Title: Effectiveness of the Routine Use of Extubation Protocol on the Incidence of Occurrence of Failures Number of Extubation in Pediatric Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6360
Record Dates: First submitted 2016-06-17; First posted 2017-04-26 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2016-05

CONDITIONS: Respiratory Insufficiency
Keywords: extubation; pediatric resuscitation; reintubation; failures of extubation.
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The failure of extubation in pediatric resuscitation is most often described as the need for reintubation within 48 hours after extubation. The failure rate of extubation in pediatric intensive care varies in the literature there is between 4 and 22% failures. These failures result in increased mortality, morbidity with a use of larger tracheostomy, a prolonged residence time. The extubation is codified in adult resuscitation and tends to be increasingly in pediatric resuscitation. In the pediatric intensive care unit of Hautepierre, a extubation protocol already exists for some time, and was prepared to go. the current literature data. It allows the harmonization of practices in service (previously left to the discretion of each doctor).

The investigators are looking to see if the protocol used systematically in the service enables a reduction in the incidence of occurrence of failures of extubation.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized in pediatric intensive care, under 18 years, intubated, ventilated for more than 2 hours and for which planning extubation or intubated children for whom an unplanned extubation just happened.
* Children whose holding parental authority are not opposed to the use of clinical data from their child for research purposes.

Exclusion Criteria:

* Refusal to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children hospitalized in pediatric intensive care, under 18 years, intubated, ventilated for more than 2 hours and for which planning extubation or intubated children for whom an unplanned extubation just happened.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Failure of extubation | need for a new intubation within the first 48 hours after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Reanimation Pediatrique Specialisee - S. Continue, Strasbourg, F, France

IPD SHARING:
Plan to Share IPD: No